CLINICAL TRIAL: NCT06430073
Title: Effect of Infections and Global DNA Methylation on Frailty Trajectories in Hospitalized Older Patients: a Multicenter Observational Study (INFRAGEN)
Brief Title: Effect of Infections and Global DNA Methylation on Frailty Trajectories in Hospitalized Older Patients (INFRAGEN)
Acronym: INFRAGEN
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Azienda Ospedaliera di Padova (Other); Fondazione IRCCS San Gerardo dei Tintori (Other); Azienda Ospedaliera Universitaria Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 83/2023/Oss/AOUFe
Record Dates: First submitted 2024-03-26; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-03

CONDITIONS: Aging; Frailty; Telomere Shortening; Inflammation; Hospital Infection
MeSH Terms: conditions — Frailty; Inflammation; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total sample: The study cohort will be composed of 340 older patients hospitalized in a Geriatric Unit with no or mild frailty in the pre-admission period, and who will present acute infections at admission or during the hospital stay.

SUMMARY:
This prospective multicenter study aims at exploring the impact of infections on intra-hospital and 3-month changes in the frailty profile of older inpatients.

To understand the complex pathways under the relationship between infections and frailty, this study will evaluate infection-related clinical and biochemical markers of systemic inflammation and genetics/epigenetics markers at ward admission.

The interplay between clinical, functional, and genetics/epigenetics factors will be evaluated in a subgroup of patients by testing whether 3-month changes in frailty concur with changes in the genomic DNA markers. This study will help characterize the pathophysiological mechanisms of frailty and identify at-risk conditions that may accelerate its course.

DETAILED DESCRIPTION:
Infectious diseases are among the most common causes of hospitalization in older adults. Indeed, recent data report that more than 15% of hospital admissions in adults 65 years or older are due to infections, mainly in the urinary and respiratory tracts. Frailty is a well-known geriatric syndrome characterized by reduced individual resilience and increased vulnerability to external stressors. The prevalence of frailty ranges from around 10% in the community setting to almost 50% among institutionalized individuals.

Although both infectious diseases and frailty are associated with negative outcomes for the health of older adults and the healthcare system, their interplay has not been largely explored. In particular, it is not clear whether and to which extent acute infectious diseases might affect frailty, fastening its development or hampering its reversion.

The overall goal of the proposed project is to evaluate the impact of acute infections on frailty trajectories in older hospitalized patients from the pre-admission status to 3 months after hospital discharge. Moreover, a comprehensive set of sociodemographic, clinical, functional, and genetic/epigenetic factors will be assessed as possible effect modifiers in the association between infections and frailty trajectories.

This multicenter prospective observational study includes four geriatric wards (Ferrara, Padova, Milano, and Napoli) and involves individuals with no or mild-to-moderate frailty. A novel and interesting aspect will be represented by the analysis of genetic and epigenetic factors, i.e. global DNA methylation and telomere length. This point will make possible exploring the complex pathophysiologic mechanisms of frailty development using a translational approach involving both basic science and clinical researchers.

Overall, this study will help better identify at-risk conditions that may accelerate the course of frailty. Therefore, the project findings may promote the importance of interventions that could counteract frailty development during the hospital stay and should be addressed primarily to the categories of patients at highest risk.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of acute infection diseases at hospital admission or during the hospital stay, according to specific ICD-9 codes with or without systemic inflammatory reaction;
* pre-admission non-frailty or mild frailty assessed using the Clinical Frailty Scale (CFS < 6).

Exclusion Criteria:

* terminally ill patients with an estimated life expectancy less than 3 months;
* presence of pre-admission frailty (CFS ≥ 6);
* unwillingness to participate in the study or to complete the follow-up assessments

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The project will involve older patients hospitalized in the Geriatric Units of the University Hospital of Ferrara, Padua, Monza, and Napoli. All patients non-frail or with mild frailty in the pre-admission period, and who will present a confirmed diagnosis of acute infection diseases at hospital admission or during the hospital stay, will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in frailty index from pre-admission to hospital discharge | From 14 days before admission to hospital discharge (up to 60 days)
  Frailty will be valuated through the Frailty Index (i.e. score from 0 to 1, with higher values corresponding to higher frailty), considering clinical and functional data. Pre-admission frailty will be retrospectively assessed to reflect the participant's status in the two weeks prior to the hospital admission. Frailty assessment will be repeated within 48h before the hospital discharge.

SECONDARY OUTCOMES:
Change in Clinical Frailty Scale from pre-admission to hospital discharge | From 14 days before admission to hospital discharge (up to 60 days)
  Frailty will be evaluated through the Clinical Frailty Scale (i.e. score from 1 to 9, with higher values corresponding to higher frailty). Pre-admission frailty will be retrospectively assessed to reflect the participant's status in the two weeks prior to the hospital admission. Frailty assessment will be repeated within 48h before the hospital discharge.
Difference in in-hospital mortality between inpatients with vs without infections with systemic inflammation | From 14 days before admission to hospital discharge (up to 60 days)
  All-cause mortality will be computed for participants with vs without infections associated with a systemic inflammatory response.
Difference in the length of hospital stay between inpatients with vs without infections with systemic inflammation | From 14 days before admission to hospital discharge (up to 60 days)
  The length of hospital stay (number of days from hospital admission to hospital discharge) will be computed for participants with vs without infections associated with a systemic inflammatory response.
Difference in the global DNA methylation between individuals with stable vs worsened frailty during the hospital stay. | From 14 days before admission to hospital discharge (up to 60 days)
  DNA extraction from whole blood will be performed by Automated Genomic DNA Purification EZ1 XL machine (QIAGEN). Global DNA methylation assessment will be performed by "highly quantitative pyrosequencing" technique as genome-wide DNA methylation levels and as gene promoter associated CpG islands utilizing selected age-related methylation marker loci and at LINE-1 repetitive elements (as a surrogate for genome-wide methylation). The patterns of global DNA methylation will be assessed in duplicate for each sample and expressed in percentage as the mean obtained by the two evaluations and considered valuable with a discrepancy <2%. Methylation percentages can be stratified into quartiles, and the middle two quartiles combined will be used as the reference category. The frequencies of individuals belonging to the highest and lowest DNA methylation quartiles will be compared between individuals reporting worsening in FI or CFS during the hospitalization vs those stable in frailty levels.
Difference in telomere length between individuals with stable vs worsened frailty during the hospital stay | From 14 days before admission to hospital discharge (up to 60 days)
  Telomere length will be compared between individuals with stable vs worsened frailty during the hospital stay. DNA extraction from whole blood will be performed by Automated Genomic DNA Purification EZ1 XL machine (QIAGEN). Leukocyte Telomere Length (LTL) will be assessed by quantitative PCR as previously described as predictors of biological age in frailty and mortality association studies. As a measure of the relative Telomere length, the ratio of the telomere repeat copy number to the number of single-copy gene ratio (T/S ratio) will be determined by quantitative PCR using the single-copy gene 36B4 for reference and a standard curve. Quality controls and assay validation tests will be assessed by official commercial recognized standards (Qiagen, LifeTechnology).
Change in frailty index from hospital discharge to 3-month follow-up | From hospital discharge until 3 months after hospital discharge (time frame: 3 months)
  Frailty will be valuated through the Frailty Index (i.e. score from 0 to 1, with higher values corresponding to higher frailty), considering clinical and functional data. Frailty assessment will be performed within 48h before the hospital discharge and after 3-month from the hospital discharge.
Change in Clinical Frailty Scale from hospital discharge to 3-month follow-up | From hospital discharge until 3 months after hospital discharge (time frame: 3 months)
  Frailty will be evaluated through the Clinical Frailty Scale (i.e. score from 1 to 9, with higher values corresponding to higher frailty). Frailty assessment will be performed within 48h before the hospital discharge and after 3-month from the hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Volpato, MD, Principal Investigator — Università degli Studi di Ferrara

REFERENCES:
- [Background] Franceschi C, Campisi J. Chronic inflammation (inflammaging) and its potential contribution to age-associated diseases. J Gerontol A Biol Sci Med Sci. 2014 Jun;69 Suppl 1:S4-9. doi: 10.1093/gerona/glu057. PMID 24833586
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Greco GI, Noale M, Trevisan C, Zatti G, Dalla Pozza M, Lazzarin M, Haxhiaj L, Ramon R, Imoscopi A, Bellon S, Maggi S, Sergi G. Increase in Frailty in Nursing Home Survivors of Coronavirus Disease 2019: Comparison With Noninfected Residents. J Am Med Dir Assoc. 2021 May;22(5):943-947.e3. doi: 10.1016/j.jamda.2021.02.019. Epub 2021 Feb 22. PMID 33757725
- [Background] Huoman J, Sayyab S, Apostolou E, Karlsson L, Porcile L, Rizwan M, Sharma S, Das J, Rosen A, Lerm M. Epigenetic rewiring of pathways related to odour perception in immune cells exposed to SARS-CoV-2 in vivo and in vitro. Epigenetics. 2022 Dec;17(13):1875-1891. doi: 10.1080/15592294.2022.2089471. Epub 2022 Jun 26. PMID 35758003
- [Background] Iwai-Saito K, Shobugawa Y, Aida J, Kondo K. Frailty is associated with susceptibility and severity of pneumonia in older adults (A JAGES multilevel cross-sectional study). Sci Rep. 2021 Apr 12;11(1):7966. doi: 10.1038/s41598-021-86854-3. PMID 33846416
- [Background] Lapham K, Kvale MN, Lin J, Connell S, Croen LA, Dispensa BP, Fang L, Hesselson S, Hoffmann TJ, Iribarren C, Jorgenson E, Kushi LH, Ludwig D, Matsuguchi T, McGuire WB, Miles S, Quesenberry CP Jr, Rowell S, Sadler M, Sakoda LC, Smethurst D, Somkin CP, Van Den Eeden SK, Walter L, Whitmer RA, Kwok PY, Risch N, Schaefer C, Blackburn EH. Automated Assay of Telomere Length Measurement and Informatics for 100,000 Subjects in the Genetic Epidemiology Research on Adult Health and Aging (GERA) Cohort. Genetics. 2015 Aug;200(4):1061-72. doi: 10.1534/genetics.115.178624. Epub 2015 Jun 19. PMID 26092717
- [Background] Park CM, Kim W, Rhim HC, Lee ES, Kim JH, Cho KH, Kim DH. Frailty and hospitalization-associated disability after pneumonia: A prospective cohort study. BMC Geriatr. 2021 Feb 5;21(1):111. doi: 10.1186/s12877-021-02049-5. PMID 33546614
- [Background] Prampart S, Le Gentil S, Bureau ML, Macchi C, Leroux C, Chapelet G, de Decker L, Rouaud A, Boureau AS. Functional decline, long term symptoms and course of frailty at 3-months follow-up in COVID-19 older survivors, a prospective observational cohort study. BMC Geriatr. 2022 Jun 30;22(1):542. doi: 10.1186/s12877-022-03197-y. PMID 35768781
- [Background] Rockwood K, Mitnitski A. Frailty in relation to the accumulation of deficits. J Gerontol A Biol Sci Med Sci. 2007 Jul;62(7):722-7. doi: 10.1093/gerona/62.7.722. PMID 17634318
- [Background] Schneider CV, Schneider KM, Teumer A, Rudolph KL, Hartmann D, Rader DJ, Strnad P. Association of Telomere Length With Risk of Disease and Mortality. JAMA Intern Med. 2022 Mar 1;182(3):291-300. doi: 10.1001/jamainternmed.2021.7804. PMID 35040871
- [Background] Schork NJ, Beaulieu-Jones B, Liang W, Smalley S, Goetz LH. Does Modulation of an Epigenetic Clock Define a Geroprotector? Adv Geriatr Med Res. 2022;4(1):e220002. doi: 10.20900/agmr20220002. Epub 2022 Mar 29. PMID 35466328
- [Background] Seligman BJ, Berry SD, Lipsitz LA, Travison TG, Kiel DP. Epigenetic Age Acceleration and Change in Frailty in MOBILIZE Boston. J Gerontol A Biol Sci Med Sci. 2022 Sep 1;77(9):1760-1765. doi: 10.1093/gerona/glac019. PMID 35037036
- [Background] Vetter VM, Kalies CH, Sommerer Y, Spira D, Drewelies J, Regitz-Zagrosek V, Bertram L, Gerstorf D, Demuth I. Relationship Between 5 Epigenetic Clocks, Telomere Length, and Functional Capacity Assessed in Older Adults: Cross-Sectional and Longitudinal Analyses. J Gerontol A Biol Sci Med Sci. 2022 Sep 1;77(9):1724-1733. doi: 10.1093/gerona/glab381. PMID 35032170
- [Background] Vlachogiannis NI, Baker KF, Georgiopoulos G, Lazaridis C, Schim van der Loeff I, Hanrath AT, Sopova K, Tual-Chalot S, Gatsiou A, Spyridopoulos I, Stamatelopoulos K, Duncan CJA, Stellos K. Clinical frailty, and not features of acute infection, is associated with late mortality in COVID-19: a retrospective cohort study. J Cachexia Sarcopenia Muscle. 2022 Jun;13(3):1502-1513. doi: 10.1002/jcsm.12966. Epub 2022 Mar 7. PMID 35257497
- [Background] Wang J, Maxwell CA, Yu F. Biological Processes and Biomarkers Related to Frailty in Older Adults: A State-of-the-Science Literature Review. Biol Res Nurs. 2019 Jan;21(1):80-106. doi: 10.1177/1099800418798047. Epub 2018 Sep 9. PMID 30198309
- [Background] Yoshikawa TT, Norman DC. Geriatric Infectious Diseases: Current Concepts on Diagnosis and Management. J Am Geriatr Soc. 2017 Mar;65(3):631-641. doi: 10.1111/jgs.14731. Epub 2017 Jan 31. PMID 28140454
- [Derived] Guo W, Bencivenga L, Zanforlini BM, Curreri C, Ferrara MC, Maisano B, Tinelli L, Ceparano LA, Merenda R, Cosma C, Manfron L, Gentili N, Sturani S, Cardi M, Campion A, Berardi B, Lombardi M, D'Aversa E, Salvatori F, Tisato V, Vargas JV, Femminella GD, Gemmati D, Sergi G, Bellelli G, Mazzola P, Trevisan C, Volpato S; INFRAGEN working group. Effect of infections, DNA methylation and telomere length on frailty trajectories in hospitalized older patients: the INFRAGEN study protocol. BMC Geriatr. 2025 Jul 23;25(1):545. doi: 10.1186/s12877-025-06194-z. PMID 40702442